CLINICAL TRIAL: NCT04679558
Title: Antibacterial Effect of Chlorhexidine Added to the Preventive Protocol in Adolescent Special Needs
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Katreen Tawfik, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7all
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Caries
MeSH Terms: interventions — Paint

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): Preventive protocol
  Interventions: Behavioral: Preventive protocol
- Intervention (Experimental): Adding chlorhexidine to the preventive protocol
  Interventions: Drug: Chlorhexidine varnish added to the preventive protocol

INTERVENTIONS:
Drug: Chlorhexidine varnish added to the preventive protocol — Antibacterial agent varnish added to the preventive protocol
  Other Names: Varnish
  Arms: Intervention
Behavioral: Preventive protocol — Preventive protocol
  Other Names: Caries preventive protocol
  Arms: Comparator

SUMMARY:
This study ia conducted to know the antibacterial effect of chlorhexidine on the mouth flora speciallly in adolescent special needs who can't hold the tooth brush properly

DETAILED DESCRIPTION:
This study ia conducted to know the antibacterial effect of chlorhexidine on the mouth flora speciallly in adolescent special needs who can't hold the tooth brush properly cause those have alot of problems concerning the accumulagio. Of plaque and so increased bacteria

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of disability like special needs autism and down syndrome

Exclusion Criteria:

* age below 13

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Streptococcus mutans count | 1 year
  Antibacterial effect of chlorhexidine on streptococcus mutans count

CONTACTS AND LOCATIONS:
Overall Officials: Katreen Fouad, Principal Investigator — Resident
Locations (1):
- School, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Journal
Supporting Information: Study Protocol
Time Frame: 10 months
Access Criteria: Journal article